CLINICAL TRIAL: NCT04783181
Title: A Phase 1/2, First-in-Human, Open-Label, Dose-Escalation Study of the Safety and Efficacy of Gene Therapy for Congenital Adrenal Hyperplasia Through Administration of an Adeno-Associated Virus (AAV) Serotype 5-Based Recombinant Vector Encoding the Human CYP21A2 Gene
Brief Title: A Study of Gene Therapy for Classic Congenital Adrenal Hyperplasia (CAH)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adrenas Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAH-301
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: CAH; Gene therapy; AAV; AAV5
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Intervention Model Description: Participants will be assigned sequentially to one of 4 dose levels depending on the date of determination of eligibility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Experimental): BBP-631 lowest dose, administered once, intravenously (IV)
  Interventions: Biological: AAV BBP-631
- Dose Level 2 (Experimental): BBP-631 middle dose, administered once, IV
  Interventions: Biological: AAV BBP-631
- Dose Level 3 (Experimental): BBP-631, high dose, administered once, IV
  Interventions: Biological: AAV BBP-631
- Dose Level 4 (Experimental): BBP-631, highest dose, administered once, IV
  Interventions: Biological: AAV BBP-631

INTERVENTIONS:
Biological: AAV BBP-631 — intravenous

SUMMARY:
This study is designed to evaluate the safety, tolerability, and efficacy of AAV5 based BBP-631 in adult participants diagnosed with classic congenital adrenal hyperplasia.

DETAILED DESCRIPTION:
Participants will receive a single dose of AAV5 based intravenous (IV) BBP-631 and will be followed for safety and efficacy for at least 5 years after the date of treatment with BBP-631.

ELIGIBILITY:
Key Inclusion Criteria

1. Adult male and non-pregnant females with classic CAH (simple virilizing or salt-wasting) due to 21-OHD
2. Screening/baseline 17-OHP levels > 5-10 × ULN and < 40 × ULN (upper limit of normal)
3. Stable oral hydrocortisone (HC) regimen as the only glucocorticoid (GC) maintenance therapy
4. Naïve to prior gene therapy or AAV-mediated therapy

Key Exclusion Criteria

1. Positive for anti-AAV5 (Adeno-Associated Virus Type 5) antibodies
2. History of adrenalectomy and/or significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events that Led to Study Discontinuation | up to 5 years
To select the optimum dose or dose range of BBP 631 for future studies | up to 5 years

SECONDARY OUTCOMES:
Change from Baseline in 17-OHP (hydroxyprogesterone) levels | Baseline, Week 52 and through study completion, an average of 5 years
Change from Baseline in androstenedione (A4) levels | Baseline, Week 52 and through study completion, an average of 5 years
Change from Baseline in endogenous cortisol levels | Baseline, Week 52 and through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Lucas Research, Inc., Morehead City, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Adrenas Therapeutics Website — https://adrenastx.com
- See also: CAH Gene Therapy Website — https://cahgenetherapy.com